CLINICAL TRIAL: NCT02864550
Title: A Randomized, Placebo-controlled Trial of Oral Doxycycline for the Prevention of Syphilis in HIV-positive Men Who Have Sex with Men (MSM)
Brief Title: Oral Doxycycline for the Prevention of Syphilis in Men Who Have Sex with Men (DaDHS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: British Columbia Centre for Disease Control (Other Government)
Responsible Party: Principal Investigator, Jonathan Troy Grennan, Physician Lead, HIV/STI program, BCCDC, British Columbia Centre for Disease Control
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BritishCCDC2
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Syphilis; Sexually Transmitted Infections
Keywords: Men who have sex with men; Human immunodeficiency virus; Doxycycline; Tetracycline
MeSH Terms: conditions — Syphilis; Sexually Transmitted Diseases; Homosexuality; Acquired Immunodeficiency Syndrome | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doxycycline arm (Experimental): Participants in this intervention group will receive doxycycline 100mg orally daily, which is available as a 100mg capsule. This single daily dose was chosen to maximize adherence, given the common use of once-daily Human Immunodeficiency Virus (HIV) pre-exposure prophylaxis (PrEP), as well as its efficacy as once-daily prophylaxis against malaria and its utility as dosing as infrequent as once weekly for another spirochete infection, leptospirosis.
  Interventions: Drug: Doxycycline
- Placebo arm (Placebo Comparator): Participants in this control group will receive a placebo capsule identical in appearance, taste, and size to the capsule provided to the intervention group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Doxycycline — doxycycline 100mg orally daily
  Arms: Doxycycline arm
Other: Placebo — placebo capsule identical in appearance, taste, and size to the capsule provided to the intervention group
  Arms: Placebo arm

SUMMARY:
Syphilis is a sexually transmitted infection (STI) disproportionately affecting gay, bisexual and other men who have sex with men (gbMSM), with the potential for significant sequelae - particularly in those who are Human Immunodeficiency Virus (HIV)-positive. Rising rates of this STI have prompted a search for novel prevention solutions. A recent pilot study of daily doxycycline prophylaxis demonstrated promise as a novel STI prevention tool. This innovative approach to STI prevention has solid clinical precedent, both from the HIV pre-exposure prophylaxis (PrEP) literature, as well as doxycycline's use as prophylaxis for other infections. The overarching goal of this project is to determine whether the daily use of doxycycline is an efficacious and acceptable intervention for syphilis prevention in high-risk, HIV-positive gbMSM.

DETAILED DESCRIPTION:
Syphilis disproportionately impacts gbMSM:

Syphilis remains an important cause of morbidity in gbMSM. Up to 75% of early syphilis infections occur in gbMSM - a population with syphilis rates nearly 10-fold higher than in those who are HIV negative. In Canada's urban centres, 2/3 of syphilis cases are in HIV-positive gbMSM, and re-infection remains high. HIV co-infection with syphilis has important implications for HIV management. Syphilis may increase HIV viral load levels in virologically suppressed individuals, and genital ulcers increase the risk of HIV transmission and acquisition.

The era of novel, biomedical prevention technologies:

Significant advancements have shaped the past two decades of HIV care. Antiretroviral therapy (ART) has substantially reduced HIV-associated morbidity and mortality and extended life expectancy to near-normal levels. With reduced morbidity and mortality associated with HIV, gbMSM may also be changing their sexual behaviours. Seroadaptive strategies, such as serosorting (selecting sexual partners of the same serostatus) and seropositioning (selecting a sexual position to minimize the risk of HIV transmission) are common among gbMSM. While this may be mitigating the risk of HIV transmission or acquisition, there is evidence to suggest that decreasing condom use may contribute to a rise in syphilis and other bacterial STIs in high-risk populations. Further, new evidence has emerged demonstrating the efficacy of HIV PrEP in preventing HIV acquisition. The combination use of tenofovir/emtricitabine was shown in the Pre-exposure Prophylaxis Initiative (iPREX) trial to reduce the risk of HIV acquisition by 44% in HIV-negative gbMSM when taken daily as PrEP. Among those with detectable drug levels, the risk reduction was > 90%.

A role for PrEP in other STIs? The exciting developments in HIV prevention have encouraged investigators to expand this strategy to the prevention of other STIs, a modality previously shown to be acceptable to gbMSM. A recent pilot study randomized participants to receive either the antimicrobial doxycycline daily or a monetary incentive to remain STI-free throughout the study period. After 48 weeks, those receiving doxycycline were significantly less likely to be diagnosed with any STI (odds ratio: 0.27; 95% confidence interval: 0.09-0.83). Though there was also a trend toward benefit for doxycycline in specifically preventing syphilis, significance was not achieved for this outcome.

The first large-scale syphilis PrEP study:

Given the rising rates of syphilis and its disproportionate impact on HIV-positive gbMSM, there is an urgent need to replicate this study on a broader scale. This proposed study will contribute to this field by being - to the investigators' knowledge - the first large-scale, methodologically rigorous trial of syphilis PrEP, and has the potential to provide a completely novel and innovative tool to the syphilis prevention armamentarium. It will provide insight on whether daily doxycycline is an efficacious PrEP intervention for the prevention of syphilis and other bacterial STIs, as well as shedding light on issues relating to its feasibility as a prevention tool, including its safety, tolerability, how well individuals adhere to it, and its impact on the development of antimicrobial resistance. These outcomes are directly in line with the planned outputs of this study, and have the potential to drastically shift how people think about and manage syphilis and other STI prevention in gbMSM.

Primary objective

1. To assess feasibility of using daily doxycycline PrEP, as defined by:

   a. Evaluation of feasibility of recruitment for a larger study i. Proportion of participants approached for study who are eligible and agree to participate.

   b. Adherence to 24 and 48 weeks of study drug (doxycycline or placebo) i. Determine proportion of individuals with >95% adherence to study drug over 24 and 48 weeks ii. Proportion of individuals in the doxycycline arm with therapeutic doxycycline plasma level at each study visit.

   c. Tolerability of doxycycline i. Comparison of grade 3 or 4 adverse events in those receiving doxycycline vs. placebo ii. Comparison of the proportion of individuals with adverse event-related discontinuation of study drug in each arm

   2.2 Secondary objectives
2. To evaluate antimicrobial resistance over time.

   a. Change in proportion of participants with evidence of tetracycline class resistance in common flora, namely Staphylococcus aureus, Streptococcus pyogenes and Streptococcus pneumoniae from baseline to 24 and 48 weeks.
3. To evaluate changes in sexual activity reported by study participants over the study period.
4. To compare syphilis incidence between those in the doxycycline vs. placebo arms.
5. To describe frequency of other STIs diagnosed in study participants over the study period.

   Exploratory objectives will include:
6. To changes in the rectal microbiome of study participants from baseline to 24 and 48 weeks after initiation of doxycycline.

ELIGIBILITY:
The inclusion criteria for this study are as follows:

1. Males, ≥ 18 years of age at baseline;
2. Self-reported MSM status;
3. Self-report condomless anal sex with a man within the last 6 months;
4. Laboratory documentation of HIV-1 infection;
5. Prior diagnosis of early/infectious syphilis (i.e. primary, secondary or early latent) within preceding 36 months (defined on the basis of a new positive serum rapid plasma reagin (RPR) test, or ≥2-dilution rise in titre if previous syphilis, or positive darkfield microscopy result or T. pallidum direct fluorescent antibody test or PCR from a primary lesion);
6. Able to provide informed consent.

The exclusion criteria for this study are as follows:

1. Known allergy or intolerance to doxycycline or tetracyclines;
2. A known diagnosis of myasthenia gravis;
3. Use of medications which could lower doxycycline levels, including barbiturates, phenytoin and carbamazepine;
4. Individuals using isotretinoin;
5. Any individual capable of getting pregnant.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
To assess the proportion of participants who are eligible and consent to participate amongst those approached. | 15 months
  To determine the feasibility of daily syphilis PrEP
To assess the proportion of participants reporting > 95% adherence to study drug, according to self-report and pill counts. | 15 months
  To determine the feasibility of daily syphilis PrEP
To assess the proportion of individuals with therapeutic doxycycline drug level (defined at ≥ 1000 ng/mL) at each study time point. | 15 months
  To determine the feasibility of daily syphilis PrEP
To assess the proportion of individuals reporting grade 3 or 4 adverse events in each study arm. | 15 months
  To determine the feasibility of daily syphilis PrEP
Proportion of individuals with adverse event-related study drug discontinuation in each study arm. | 15 months
  To determine the feasibility of daily syphilis PrEP

SECONDARY OUTCOMES:
To assess the proportion of individuals with evidence of tetracycline class resistance in common flora (Staphylococcus aureus, Streptococcus pyogene and Streptococcus pneumoniae) | At 6 and 12 months
  To evaluate tetracycline class resistance in common flora (i.e. syphilis, gonorrhea, or chlamydia)
To assess the changes in sexual risk behaviour will be calculated by comparing risk parameters (i.e. number partners, number of anal sexual encounters that were condomless) from pre-PrEP initiation to the study period. | 15 months
  Change in sexual behaviour will also be compared between study arms.
To assess the incidence of early syphilis infection | 15 months
  To evaluate syphilis and other STI incidence over the study period.
To assess the incidence of gonorrhea or chlamydia infection | 15 months
  To evaluate syphilis and other STI incidence over the study period.

OTHER OUTCOMES:
To assess changes in the bacterial populations found in the rectal microbiome. | 15 months
  Exploratory outcome: to assess % changes of each bacterial genus in rectal microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Troy Grennan, MD, Principal Investigator — BC Centre for Disease Control
Locations (1):
- British Columbia Centre for Disease Control, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ontario Agency for Health Protection and Promotion (Public Health Ontario). Reportable Disease Trends in Ontario, 2013. Toronto, ON: Queen's Printer for Ontario; 2015.
- [Background] Burchell AN, Allen VG, Gardner SL, Moravan V, Tan DH, Grewal R, Raboud J, Bayoumi AM, Kaul R, Mazzulli T, McGee F, Rourke SB; OHTN Cohort Study Team. High incidence of diagnosis with syphilis co-infection among men who have sex with men in an HIV cohort in Ontario, Canada. BMC Infect Dis. 2015 Aug 20;15:356. doi: 10.1186/s12879-015-1098-2. PMID 26289937
- [Background] Bolan RK, Beymer MR, Weiss RE, Flynn RP, Leibowitz AA, Klausner JD. Doxycycline prophylaxis to reduce incident syphilis among HIV-infected men who have sex with men who continue to engage in high-risk sex: a randomized, controlled pilot study. Sex Transm Dis. 2015 Feb;42(2):98-103. doi: 10.1097/OLQ.0000000000000216. PMID 25585069
- [Background] Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV; iPrEx Study Team. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med. 2010 Dec 30;363(27):2587-99. doi: 10.1056/NEJMoa1011205. Epub 2010 Nov 23. PMID 21091279
- [Background] Grant RM, Anderson PL, McMahan V, Liu A, Amico KR, Mehrotra M, Hosek S, Mosquera C, Casapia M, Montoya O, Buchbinder S, Veloso VG, Mayer K, Chariyalertsak S, Bekker LG, Kallas EG, Schechter M, Guanira J, Bushman L, Burns DN, Rooney JF, Glidden DV; iPrEx study team. Uptake of pre-exposure prophylaxis, sexual practices, and HIV incidence in men and transgender women who have sex with men: a cohort study. Lancet Infect Dis. 2014 Sep;14(9):820-9. doi: 10.1016/S1473-3099(14)70847-3. Epub 2014 Jul 22. PMID 25065857
- [Background] Pang LW, Limsomwong N, Boudreau EF, Singharaj P. Doxycycline prophylaxis for falciparum malaria. Lancet. 1987 May 23;1(8543):1161-4. doi: 10.1016/s0140-6736(87)92141-6. PMID 2883488
- [Background] Sehgal SC, Sugunan AP, Murhekar MV, Sharma S, Vijayachari P. Randomized controlled trial of doxycycline prophylaxis against leptospirosis in an endemic area. Int J Antimicrob Agents. 2000 Feb;13(4):249-55. doi: 10.1016/s0924-8579(99)00134-x. PMID 10755239
- [Background] Patton ME, Su JR, Nelson R, Weinstock H; Centers for Disease Control and Prevention (CDC). Primary and secondary syphilis--United States, 2005-2013. MMWR Morb Mortal Wkly Rep. 2014 May 9;63(18):402-6. PMID 24807239
- [Background] Jin F, Prestage GP, Zablotska I, Rawstorne P, Imrie J, Kippax SC, Donovan B, Templeton DJ, Kaldor JM, Grulich AE. High incidence of syphilis in HIV-positive homosexual men: data from two community-based cohort studies. Sex Health. 2009 Dec;6(4):281-4. doi: 10.1071/SH09060. PMID 19917195
- [Background] Ling DI, Janjua NZ, Wong S, Krajden M, Hoang L, Morshed M, Achen M, Murti M, Lester RT, Wong J, Ogilvie G, Gilbert M. Sexually transmitted infection trends among gay or bisexual men from a clinic-based sentinel surveillance system in British Columbia, Canada. Sex Transm Dis. 2015 Mar;42(3):153-9. doi: 10.1097/OLQ.0000000000000250. PMID 25668648
- [Background] Ogilvie GS, Taylor DL, Moniruzzaman A, Knowles L, Jones H, Kim PH, Rekart ML. A population-based study of infectious syphilis rediagnosis in British Columbia, 1995-2005. Clin Infect Dis. 2009 Jun 1;48(11):1554-8. doi: 10.1086/598997. PMID 19402790
- [Background] Jarzebowski W, Caumes E, Dupin N, Farhi D, Lascaux AS, Piketty C, de Truchis P, Bouldouyre MA, Derradji O, Pacanowski J, Costagliola D, Grabar S; FHDH-ANRS CO4 Study Team. Effect of early syphilis infection on plasma viral load and CD4 cell count in human immunodeficiency virus-infected men: results from the FHDH-ANRS CO4 cohort. Arch Intern Med. 2012 Sep 10;172(16):1237-43. doi: 10.1001/archinternmed.2012.2706. PMID 22826097
- [Background] Fleming DT, Wasserheit JN. From epidemiological synergy to public health policy and practice: the contribution of other sexually transmitted diseases to sexual transmission of HIV infection. Sex Transm Infect. 1999 Feb;75(1):3-17. doi: 10.1136/sti.75.1.3. PMID 10448335
- [Background] Palella FJ Jr, Delaney KM, Moorman AC, Loveless MO, Fuhrer J, Satten GA, Aschman DJ, Holmberg SD. Declining morbidity and mortality among patients with advanced human immunodeficiency virus infection. HIV Outpatient Study Investigators. N Engl J Med. 1998 Mar 26;338(13):853-60. doi: 10.1056/NEJM199803263381301. PMID 9516219
- [Background] Lohse N, Hansen AB, Pedersen G, Kronborg G, Gerstoft J, Sorensen HT, Vaeth M, Obel N. Survival of persons with and without HIV infection in Denmark, 1995-2005. Ann Intern Med. 2007 Jan 16;146(2):87-95. doi: 10.7326/0003-4819-146-2-200701160-00003. PMID 17227932
- [Background] Samji H, Cescon A, Hogg RS, Modur SP, Althoff KN, Buchacz K, Burchell AN, Cohen M, Gebo KA, Gill MJ, Justice A, Kirk G, Klein MB, Korthuis PT, Martin J, Napravnik S, Rourke SB, Sterling TR, Silverberg MJ, Deeks S, Jacobson LP, Bosch RJ, Kitahata MM, Goedert JJ, Moore R, Gange SJ; North American AIDS Cohort Collaboration on Research and Design (NA-ACCORD) of IeDEA. Closing the gap: increases in life expectancy among treated HIV-positive individuals in the United States and Canada. PLoS One. 2013 Dec 18;8(12):e81355. doi: 10.1371/journal.pone.0081355. eCollection 2013. PMID 24367482
- [Background] Bogowicz P, Moore D, Kanters S, Michelow W, Robert W, Hogg R, Gustafson R, Gilbert M; ManCount Study Team. HIV testing behaviour and use of risk reduction strategies by HIV risk category among MSM in Vancouver. Int J STD AIDS. 2016 Mar;27(4):281-7. doi: 10.1177/0956462415575424. Epub 2015 Mar 2. PMID 25736346
- [Background] Vallabhaneni S, McConnell JJ, Loeb L, Hartogensis W, Hecht FM, Grant RM, Pilcher CD. Changes in seroadaptive practices from before to after diagnosis of recent HIV infection among men who have sex with men. PLoS One. 2013;8(2):e55397. doi: 10.1371/journal.pone.0055397. Epub 2013 Feb 6. PMID 23405145
- [Background] Hart G. Syphilis tests in diagnostic and therapeutic decision making. Ann Intern Med. 1986 Mar;104(3):368-76. doi: 10.7326/0003-4819-104-3-368. PMID 3511822
- [Background] Romney MG, Hull MW, Gustafson R, Sandhu J, Champagne S, Wong T, Nematallah A, Forsting S, Daly P. Large community outbreak of Streptococcus pneumoniae serotype 5 invasive infection in an impoverished, urban population. Clin Infect Dis. 2008 Sep 15;47(6):768-74. doi: 10.1086/591128. PMID 18690803
- [Background] Lloyd-Smith E, Hull MW, Hawkins D, Champagne S, Kerr T, Romney MG. Screening for methicillin-resistant Staphylococcus aureus (MRSA) in community-recruited injection drug users: are throat swabs necessary? Epidemiol Infect. 2012 Sep;140(9):1721-4. doi: 10.1017/S0950268811002421. Epub 2011 Dec 13. PMID 22152523
- [Background] Kuehnert MJ, Kruszon-Moran D, Hill HA, McQuillan G, McAllister SK, Fosheim G, McDougal LK, Chaitram J, Jensen B, Fridkin SK, Killgore G, Tenover FC. Prevalence of Staphylococcus aureus nasal colonization in the United States, 2001-2002. J Infect Dis. 2006 Jan 15;193(2):172-9. doi: 10.1086/499632. Epub 2005 Dec 15. PMID 16362880
- [Background] Abudu L, Blair I, Fraise A, Cheng KK. Methicillin-resistant Staphylococcus aureus (MRSA): a community-based prevalence survey. Epidemiol Infect. 2001 Jun;126(3):351-6. doi: 10.1017/s0950268801005416. PMID 11467791
- [Background] Fedson DS, Scott JA. The burden of pneumococcal disease among adults in developed and developing countries: what is and is not known. Vaccine. 1999 Jul 30;17 Suppl 1:S11-8. doi: 10.1016/s0264-410x(99)00122-x. PMID 10471174
- [Background] Aral SO, Blanchard JF. The Program Science initiative: improving the planning, implementation and evaluation of HIV/STI prevention programs. Sex Transm Infect. 2012 Apr;88(3):157-9. doi: 10.1136/sextrans-2011-050389. Epub 2012 Feb 22. PMID 22363021